CLINICAL TRIAL: NCT05541081
Title: Investigating Point-of-care Diagnostics for Sexually Transmitted Infections and Antimicrobial Resistance in Primary Care in Zimbabwe
Acronym: IPSAZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Biomedical Research and Training Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 26787
Record Dates: First submitted 2022-08-23; First posted 2022-09-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Sexually Transmitted Infection; Chlamydia; Gonorrhea; Trichomoniasis; Syphilis; Hepatitis B; HIV Infections; Pregnancy; Sexually Transmitted Diseases
Keywords: Antenatal care; Sexual and reproductive healthcare; Zimbabwe
MeSH Terms: conditions — Sexually Transmitted Diseases; Chlamydia Infections; Gonorrhea; Trichomonas Infections; Syphilis; Hepatitis B; HIV Infections; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Point-of-care STI testing (Other): Provision of point-of-care testing for chlamydia, gonorrhoea, trichomoniasis, syphilis, HIV, and hepatitis B, with comprehensive case management including partner notification
  Interventions: Diagnostic Test: Point-of-care STI testing

INTERVENTIONS:
Diagnostic Test: Point-of-care STI testing — Testing for:
  * Chlamydia and gonorrhoea using the GeneXpert platform (Cepheid)
  * Trichomoniasis using the OSOM Trichomonas Rapid Test (Sekisui Diagnostics)
  * HIV and syphilis using the SD BIOLINE HIV/Syphilis Duo (Abbott Diagnostics Medical Co. Ltd)
  * Hepatitis B using the HBsAg2 rapid test (Abbott Diagnostics Medical Co. Ltd)

SUMMARY:
A prospective interventional study to evaluate a strategy of point-of-care testing for sexually transmitted infections including chlamydia, gonorrhoea, trichomoniasis, syphilis, and Hepatitis B with comprehensive case management including partner notification in antenatal settings in Harare province, Zimbabwe.

DETAILED DESCRIPTION:
Sexually transmitted infections (STIs) can cause serious morbidity including pelvic inflammatory disease, infertility, poor mental health, adverse pregnancy outcomes and an increased risk of HIV transmission. In low and middle-income countries (LMICs), STIs are treated using syndromic management, which has poor sensitivity and specificity, leading to considerable levels of both underdiagnosis and overtreatment. In recent years, simpler diagnostic platforms for STIs have been developed. Development and evaluation of strategies for provision of diagnostic testing in LMICs are needed and the World Health Organization (WHO) has called for evidence to inform replacement of syndromic management by diagnostic testing.

The aim of this project is to evaluate a strategy of point-of-care (POC) testing for STIs including chlamydia, gonorrhoea, trichomoniasis, syphilis, and Hepatitis B with comprehensive case management including partner notification in antenatal settings in Harare province, Zimbabwe.

The objectives are to:

1. Determine the uptake, prevalence and yield of chlamydia, gonorrhoea, trichomoniasis, syphilis and hepatitis B testing, and risk factors for infection among women attending for antenatal care
2. Assess the acceptability and feasibility of this intervention
3. Estimate the cost and cost-effectiveness of POC STI testing
4. Investigate the prevalence of antimicrobial resistance for Neisseria gonorrhoeae to inform the development of a gonococcal antimicrobial resistance surveillance programme
5. Assess an incentives-based approach to optimize uptake of client-referral partner notification.

A prospective interventional study will be conducted in three primary healthcare clinics (PHCs) in Harare province, Zimbabwe. 1000 pregnant women will be recruited over a nine month period when registering for routine antenatal care. Testing will be staggered across sites so that testing will be available at each site for three months within the nine-month study period. All Identified STIs will be managed comprehensively including treatment and/or referral if required according to national guidelines, and partner notification and risk reduction counselling.

Given the relatively low number of gonococcal isolates likely to be obtained from pregnant women alone, men attending the PHCs with urethral discharge will be recruited to gain sufficient numbers to establish a surveillance programme. Urethral samples will be collected from 140 men with urethral discharge, to support the assessment of antimicrobial resistance amongst patients with gonorrhoea.

ELIGIBILITY:
Inclusion criteria:

* Pregnant woman
* Attending a study site for antenatal care

Exclusion criteria:

* Enrolment in this study on a previous antenatal visit
* Unable to provide consent in English or Shona

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Composite STI prevalence | Through study completion, up to 1 year
  Composite % of participants with chlamydia, gonorrhoea, trichomoniasis, syphilis, and/or hepatitis B
Individual STI prevalences | Through study completion, up to 1 year
  Individual % of participants with chlamydia, gonorrhoea, trichomoniasis, syphilis, and hepatitis B

SECONDARY OUTCOMES:
Uptake of STI testing | Through study completion, up to 1 year
  % of individuals approached who accept and undergo testing
Yield of STI testing | Through study completion, up to 1 year
  % of individuals approached who test positive for an STI
Uptake of treatment | Through study completion, up to 1 year
  % of participants with a curable STI who accept treatment
Uptake of partner notification | Through study completion, up to 1 year
  % of participants with a curable STI who undertake partner notification
Prevalence of antimicrobial resistance in gonococcal isolates | Through study completion, up to 1 year
  % of gonococcal isolates with resistance to ceftriaxone, cefixime, azithromycin, and ciprofloxacin
Prevalence of adverse birth outcomes | Through study completion, up to 2 years
  % of pregnancies with premature birth, miscarriage, or low birth weight

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Martin, MBBS, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Mbare polyclinic, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
At the time of publication of research, the subset of data required for the purposes of verifying research findings will be made available for sharing and will be placed in Data Compass (the LSHTM institutional research data repository). This repository will enable direct download of records with codebooks to enable replication of the data analyses. A more complete sharing of data with any research group requesting access to individual data records will be done 12 months after publication. At this point, all data and study tools will be made available through Data Compass. Data for sharing will be de-identified prior to release. In addition, annotated questionnaires and STATA do-files used for data cleaning and analysis will be available. All databases will be accessible to authorised personnel only. Details of how to access data will be published with each study publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Complete data will be shared 12 months after publication
Access Criteria: If access to the data is requested for the purposes of re-analysis and publication, such access will only be granted if a Zimbabwean colleague is included in any resulting manuscripts as a collaborator and author. Data users will be required to acknowledge the source of data and to ensure that the regulatory requirements of the Medical Research Council of Zimbabwe (MRCZ) are met.

REFERENCES:
- [Derived] Martin K, Mackworth-Young CRS, Dauya E, Nyamwanza R, Dziva Chikwari C, Tshuma M, Tucker JD, Simms V, Bandason T, Ndowa F, Katsidzira L, Mugurungi O, Machiha A, Peters RPH, Marks M, Kranzer K, Ferrand RA. Integrating point-of-care screening for curable sexually transmitted infections with HIV, syphilis and hepatitis B screening in antenatal care services in Zimbabwe: a mixed-methods process evaluation. BMJ Glob Health. 2025 Dec 5;10(12):e019820. doi: 10.1136/bmjgh-2025-019820. PMID 41360480
- [Derived] Martin K, Mackworth-Young CRS, Nyamwanza R, Chikwari CD, Dauya E, Tucker JD, Simms V, Bandason T, Ndowa F, Machiha A, Bernays S, Marks M, Kranzer K, Ferrand RA. Financial incentives to improve uptake of partner treatment for sexually transmitted infections in antenatal care: a cluster randomised trial in Zimbabwe. Lancet Glob Health. 2025 Dec;13(12):e2097-e2110. doi: 10.1016/S2214-109X(25)00306-7. PMID 41240948
- [Derived] Martin K, Dziva Chikwari C, Dauya E, Mackworth-Young CRS, Bath D, Tucker J, Simms V, Bandason T, Ndowa F, Katsidzira L, Mugurungi O, Machiha A, Marks M, Kranzer K, Ferrand R. Investigating point-of-care diagnostics for sexually transmitted infections and antimicrobial resistance in antenatal care in Zimbabwe (IPSAZ): protocol for a mixed-methods study. BMJ Open. 2023 Apr 20;13(4):e070889. doi: 10.1136/bmjopen-2022-070889. PMID 37080628
- See also: The Health Research Unit Zimbabwe (THRU ZIM) — https://www.thruzim.org/
- See also: LSHTM Data Compass — http://datacompass.lshtm.ac.uk/